CLINICAL TRIAL: NCT02533661
Title: Effects of Family-Centered Intervention for Preterm Infants at Preschool Age
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 201412127RINC
Record Dates: First submitted 2015-08-18; First posted 2015-08-27 (Estimated); Last update posted 2019-03-07 (Actual); Status verified 2016-10

CONDITIONS: Premature Birth
Keywords: Effectiveness; Genes; Intervention; Neurodevelopment; Prematurity; Preschool Age
MeSH Terms: conditions — Premature Birth | interventions — Early Intervention, Educational

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Family-centered intervention program (Experimental): The FCIP group received:
  1. In-hospital intervention: modulation of the NICU, teaching of child development skills, feeding support,massage,parent support and education,transition home preparation.
  2. After-discharge: clinic (1, 2, 4, 9 months) and home visits (0, 6, 12 months) for teaching of child development skills, feeding support, dyadic interaction activities, modulations of home environment, parent support and education.
  Interventions: Other: Family-centered intervention program
- Usual care program (No Intervention): The UCP group received:
  1. In-hospital intervention: environmental modulation and teaching of child development skills.
  2. After-discharge:telephone calls (0, 1, 2, 4, 6, 9 and 12 months): consultation on general care concerns

INTERVENTIONS:
Other: Family-centered intervention program — This program will include in-hospital intervention, after-discharge intervention and neonatal follow-up. Five sessions of in-hospital intervention will emphasize modulation of the NICU, teaching of child developmental skills, feeding support, massage, interactional activities and parent support and education. The 7-session after-discharge intervention will consist of 4 clinic visits and 3 home visits with specific care in modulation of home environment, teaching of child developmental skills, feeding support, teaching of interactional activities, and parent support and education
  Other Names: early intervention program
  Arms: Family-centered intervention program

SUMMARY:
Accumulating data on early intervention for preterm infants in Western countries have demonstrated short- to medium-term benefits on enhancing child cognitive outcome. Furthermore, the cumulative plasticity of dopamine-related genes may interact with environmental intervention in influencing a child's behavior. However, rare studies have examined the long-term effect of early intervention for preterm infants in Eastern society and whether the genetic markers interact with environmental intervention in shaping child developmental outcomes. To meet the contemporary concept of family-centered intervention and to adapt the findings of our previous studies into program design, we have developed a family-centered intervention program (FCIP) for preterm infants with very low birth weight (VLBW, birth weight <1,500 g) in Taiwan and employed a multi-centered, randomized controlled study design to examine its short-term effects with respect to a usual care program (UCP) and its biosocial pathways.The FCIP contained ecologically pervasive child-, parent- and dyad-focused services that lasted from hospitalization until 12 months; the UCP contained child-focused services in hospitalization and phone calls after discharge. This three-year multi-centered study is therefore aimed to extend our research to examine the long-term effectiveness of FCIP on child and parent outcome compared to a usual care program (UCP) for VLBW preterm children in Taiwan at preschool age and to investigate if dopamine-related genes moderate intervention effect on child developmental outcome. A total of 275 ( 269 participants + 6 pilots) VLBW preterm infants have been enrolled and randomly assigned to the FCIP and UCP, and their buccal cells samples have been collected for typing of dopamine-related genes. All infants and families will be examined at 3 and 4 years of age for child and parent outcomes. Child outcomes will include growth, health, cognition, language, motor function, and behavioral measures; parent outcomes will consist of parental stress and quality of life measures. The long-term effect of early intervention for preterm infants will provide important information to help medical/educational professionals and public policy makers develop and assess effective intervention for Taiwanese preterm children who are at risk of developmental disorders. Furthermore, the results will help reveal the gene and intervention interaction on child developmental outcome.

DETAILED DESCRIPTION:
Study Purposes:

This study is to extend our previous research to longitudinally examine the effectiveness of FCIP and UCP for VLBW preterm children in Taiwan at 3 and 4 years of age and to investigate if dopamine-related genes moderate intervention effect on child developmental outcome. Effectiveness examined will include child and parent outcomes. Child outcomes will consist of growth, health, neurodevelopment (cognition, language and motor function) and behavior. Parent outcomes will include parental stress and quality of life. The long-term effect of early intervention for preterm children from the neonatal period to preschool age will provide important information to help medical professionals and public policy makers to develop effective intervention for Taiwanese preterm children who are at risk of developmental problems. Furthermore, the genetic susceptibility theory and the cumulative genetic plasticity theory will be used to examine the relations of polymorphisms of dopamine-related genes with child development and their possible interactions with environmental intervention on child development. Over twenty dopamine genetic markers that were identified in extensive research as being associated with plasticity for neurodevelopmental functions will be examined for their individual and synergistic influences on developmental outcomes.

Participants:

Two hundred and seventy-five VLBW preterm children participating in our previous study who were born or admitted at National Taiwan University Hospital (NTUH), Mackay Memorial Hospital (MMH) and National Cheng Kung University Hospital (NCKUH) during the period of April 2012 to December 2014 will be enrolled in this study.

Methods:

All families will be contacted via phone call and mail to participate in this study. Children and their parents will be examined for the following outcomes when the children approach 3 and 4 years of age. All measures will be conducted at the Infant Motor Development Laboratory, School of Physical Therapy, National Taiwan University, and the Cognitive Electrophysiology Laboratory, Institute of Cognitive Science, National Cheng Kung University. The outcome measures in this study will consist of the primary child outcome (growth, health, neurodevelopment [cognitive, language and motor function] and behavior) and the secondary parent outcome (parental stress and quality of life). Child neurodevelopment will be examined using the Bayley Scales of Infant Development- 2nd edition, Bayley Scales of Infant and Toddler Development-3rd edition, Movement Assessment Battery for Children-2nd Edition, and Wechsler PreSchool and Primary Scales of Intelligence-4th Edition. Child behavior will be examined using the Children's Behavior Questionnaire, Swanson, Nolan, and Pelham Questionnaire- 4th Edition, and Child Behavior Check List/4-18. Parental stress will be assessed using the Parenting Stress Index-Long Form and quality of life will be assessed using the Chinese Version World Health Organization Quality of Life- Brief Taiwan Version. Each assessment will be delineated as follows.

ELIGIBILITY:
The inclusion criteria for VLBW preterm infants were:

1. birth weight less than 1,500 gram
2. gestational age lower than 37 weeks

The inclusion criteria for parents were:

1. mothers older than 18 years of age;
2. Taiwan nationality
3. absence of maternal substance abuse (alcohol or drug)
4. married or living together at delivery
5. families residing in northern or southern Taiwan.

The exclusion criteria for VLBW preterm infants were:

1. congenital abnormality
2. severe neonatal and perinatal diseases: Severe neonatal diseases refer to major neurologic abnormalities (e.g., seizures, hydrocephalus, ventriculoperitoneal shunt, meningitis, periventricular leukomalacia, grade III-IV intraventricular hemorrhage and stage IV-V retinopathy of prematurity), necrotizing enterocolitis grade II and severe cardiopulmonary disease requiring daily oxygen use at hospital discharge that may require intensive developmental intervention and therefore did not suit for our interventions.

Furthermore, infants exhibiting persistently unstable physiological conditions until 36 weeks' PMA or older, being discharged from hospital at 44 weeks' PMA or older, or developing severe neonatal diseases were early terminated.

Ages: 3 Years to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 220 (Actual)
Dates: Start 2015-08; Primary Completion 2018-11-11 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Child: Health status | up to 2 years
  Chart review
Child: Growth - weight | up to 2 years
  weight will be assessed using an electric weight scale (kg)
Child: Growth - height | up to 2 years
  height will be assessed by the tape measure in standing position (cm)
Child: Growth - head circumference | up to 2 years
  head circumference will be assessed as the largest dimension around the head obtained with a type measure placed snugly above the ears (cm)
Child: Neurodevelopment - Bayley Scale of Infant and Toddler Development- 2nd and 3rd Edition | 1 year
  The BSID-II is a norm-referenced developmental diagnostic test for infants aged from 1 month to 42 months. The assessment contains the Motor Scale (111 items), the Mental Scale (178 items), and the Behavioral Rating Scale (30 items).
Child: Neurodevelopment - The Wechsler Preschool and Primary Scale of Intelligence-Revised Edition | 1 year
  The WPPSI-R measures cognitive development of children who aged from 3 to 7 years old. The test structure of WPPSIR-IV includes 12 subscales and three levels of interpretation: full intelligence quotient (FIQ); performance intelligence quotient (PIQ), and verbal intelligence quotient (VIQ).
Child: Neurodevelopment - Movement Assessment Battery for Children- 2nd Edition | 1 year
  The Movement ABC-II examines the movement performance in children aged 3 years to 16 years and 11 months. The assessment contains eight items that measure a child's performance of age-appropriate tasks in the aspects of manual dexterity, aiming and catching, and balance.
Child: Behavior - Children's Behavior Questionnaire | 1 year
  The CBQ is a parent-report temperament questionnaire for preschool- and school-aged children. A total of 195 items described children's reactions on 15 primary temperament characteristics: positive anticipation, smiling/laughter, high intensity pleasure, activity level, impulsivity, shyness, discomfort, fear, anger/frustration, sadness, soothability, inhibitory control, attentional focusing, low intensity pleasure, and perceptual sensitivity.
Child: Behavior - Swanson, Nolan, and Pelham Questionnaire, version IV | 1 year
  The SNAP-IV questionnaire examines the severity of ADHD and ODD in preschool- and school-aged children. The scale employs the direct symptom of Diagnosis and Statistical Manual of Mental Disorder-IV (DSM-IV) that consists of inattention (nine items), hyperactivity/impulsivity (nine items) of the criteria for ADHD, and the oppositional symptoms (eight items) of the criteria for ODD.
Child: Behavior - Child Behavior Check List/1.5-5 | 1 year
  The CBCL/1.5-5 is a parent-report questionnaire designed to assess the behavior problems in children at 1.5 to 5 years of age. The CBCL/1.5-5 consists of 99 items to assess concerning behavioral/emotional problems.
Child: Neurodevelopment - The Berry-Buktenica Developmental Test of Visual-Motor Integration | 1 year
  The VMI screens for visual-motor deficits in children from 2 to 18 years old and adults. The assessment contains visual-motor integration, visual perception and motor coordination.

SECONDARY OUTCOMES:
Parent: Parental stress - Parenting Stress Index/ Long Form | 1 year
  The PSI-LF is a self-report questionnaire that measures parenting stress based on interrelationship between the child's and the parents'characteristics. The questionnaire has 101 items, rated on a 5-point Likert scale, and contains parental distress (PD), parent-child dysfunctional interaction (PCDI), and difficult child (DC) subscales.
Parent: Quality of life - World Health Organization Quality of Life- Brief Taiwan Version | 1 year
  The WHOQOL-BREF-TW is a self-administered scale that examines the quality of life of an individual. Twenty eight items are grouped into general QOL and general health; 26 items are classified into physical, psychological, social relationship and environment domains. Items are scored from 1 to 5 on a Likert's scale.
Child: Neurophysiological functions | 1 year
  Child's neurophysiological functions will be measured by the cognitive task (eg. Go-Nogo task and oddball task) with electroencephalogram (EEG)/event-related potential (ERP) technique for the participating children at 4 years old.

CONTACTS AND LOCATIONS:
Overall Officials: Suh-Fang Jeng, Principal Investigator — School and Graduate Institute of Physical Therapy, College of Medicine, National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Zhongzheng District, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Li SJ, Tsao PN, Tu YK, Hsieh WS, Yao NJ, Wu YT, Jeng SF. Cognitive and motor development in preterm children from 6 to 36 months of age: Trajectories, risk factors and predictability. Early Hum Dev. 2022 Sep;172:105634. doi: 10.1016/j.earlhumdev.2022.105634. Epub 2022 Jul 28. PMID 35921693